CLINICAL TRIAL: NCT04476797
Title: GRECO-1: Phase I/II, Randomized, Placebo-Controlled Study of Stereotactic Body Radiation Therapy (SBRT) and GC4711 for Centrally Located or Large, Node-Negative Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Phase I/II Study of SBRT and GC4711 for Centrally Located or Large NSCLC
Acronym: GRECO-1
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development GC4711 was halted after the lead study in pancreatic cancer was stopped early due to meeting the requirements of a futility analysis
Sponsor: Galera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GTI-4711-101
Record Dates: First submitted 2020-07-15; First posted 2020-07-20 (Actual); Results first posted 2024-04-03 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-12

CONDITIONS: SBRT; NSCLC; Non-metastatic
Keywords: lymph node negative NSCLC; centrally located NSCLC; large NSCLC; SBRT

STUDY DESIGN:
Intervention Model Description: After the open label Phase 1 portion, subjects in the Phase2 portion will be randomized in a 1:1 ratio to receive GC4711 or placebo before each fraction of SBRT
Who Masked: Participant, Care Provider, Investigator
Masking Description: Phase 2 is a randomized, placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 1 GC4711 + SBRT (Experimental)
  Interventions: Drug: GC4711 +SBRT
- Phase 2 Placebo + SBRT (Placebo Comparator)
  Interventions: Drug: Placebo +SBRT
- Phase 2 GC4711 +SBRT (Experimental)
  Interventions: Drug: GC4711 +SBRT

INTERVENTIONS:
Drug: GC4711 +SBRT — 15 minute IV Infusion prior to SBRT
  Other Names: rucosopasem manganese
  Arms: Phase 1 GC4711 + SBRT; Phase 2 GC4711 +SBRT
Drug: Placebo +SBRT — 15 minute IV infusion prior to SBRT
  Arms: Phase 2 Placebo + SBRT

SUMMARY:
GTI-4711-101 is a Phase I/II study of the safety of GC4711, its effect on in-field tumor response and its potential to reduce radiation-related pulmonary injury due to SBRT for lymph node negative (T1 to T3N0M0) peripheral or central localized (within 2cm of the proximal bronchial tree) NSCLC.

After an open-label, Phase 1, safety cohort of 5 subjects has been completed, a randomized, placebo-controlled Phase 2 portion of 66 subjects will be conducted.

DETAILED DESCRIPTION:
Subjects must be referred for SBRT with large peripheral lesions (>1cm-7cm) and/or central localized, node negative, non-metastatic NSCLC, and have an ECOG PS score of 0-3. Feasibility of SBRT is judged by the treating physician.

SBRT is planned for the tumor location as a dose of or 3 fractions of 18-20 Gy (Phase 2 only) or 5 fractions of 10-12 Gy. SBRT fractions will be given within 180 minutes from the end of the GC4711 or placebo infusion.

After completion of Phase I, a Phase II, randomized, placebo-controlled study will be initiated, wherein approximately 66 subjects referred for SBRT with early stage large and/or central localized NSCLC will be randomized in a 1:1 ratio to receive either GC4711 or placebo given intravenously (IV) over 15 minutes before each fraction of SBRT, beginning the day of the first fraction of SBRT and ending the last day of SBRT.

Subjects will be monitored for treatment emergent adverse events for 30 days post SBRT completion. Additionally, subjects will be monitored 90 days post-SBRT for all adverse events to evaluate acute toxicities, and monitored for 1-year post-SBRT completion for specific late toxicities.

In-field tumor response and overall survival will be evaluated through 24 months post SBRT completion.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects at least 18 years of age.
2. Ability to understand and the willingness to sign a written informed consent.
3. Histological or biopsy proven NSCLC.
4. ECOG performance status of 0-3.
5. Node negative (T1 to T3N0M0), centrally located (within 2cm in all directions around the proximal bronchial tree, including ultra-central tumors, abutting the bronchial tree or trachea) or large (>1-7cm) Non-Small Cell Lung Cancer (NSCLC), judged acceptable for SBRT by the treating Investigator
6. Adequate end-organ function, based on routine clinical and laboratory workup:

   1. ANC >1,000 cells/µl, Platelets ≥ 75,000 cells/µl, Hemoglobin ≥ 7.0 g/dl
   2. Serum creatinine ≤ 2 x ULN or calculated creatinine clearance ≥ 30 ml/min
   3. Total bilirubin ≤ 1.5 x ULN (or direct bilirubin below the ULN), AST and ALT ≤ 2.5 x ULN
7. Males and females of must agree to use effective contraception starting prior to the first day of treatment and continuing after the last dose of GC4711/Placebo for 30 days (females) and 90 days (males).

Exclusion Criteria:

1. Subjects with confirmed nodal and/or distant disease(including brain), according standard workup by local investigator
2. Subjects with peripheral lesions 1cm or smaller
3. Prior treatment with immunotherapy within 3 months prior to Day 1 dosing.
4. Prior intra-thoracic radiotherapy or surgery with substantial overlap to planned radiation fields as determined by the treating radiation oncologist.
5. Subjects not recovered/controlled from prior treatment-related (chemotherapy or targeted therapy) toxicities judged by treating physician.
6. Uncontrolled malignancy other than lung cancer that requires active treatment or is deemed by the treating physicians to be likely to affect the subject's survival duration.
7. History of allergic reactions attributed to compounds of similar chemical or biologic composition to GC4711.
8. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
9. Participation in other clinical trials actively testing new anti-cancer treatments, unless previously written approval is provided by the Sponsor.
10. Requirement for concurrent treatment with nitrates or other drugs that may, in the judgment of the treating investigator, create a risk for a precipitous decrease in blood pressure.
11. Female subjects who are pregnant or breastfeeding.
12. Any other conditions that, in the Investigator's opinion, might indicate the subject to be unsuitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2020-10-18 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eugene P Kennedy, MD, Study Chair — Chief Medical Officer
Locations (10):
- United States (10):
  - Banner MD Anderson Cancer Center at NCMC, Greeley, Colorado
  - Banner McKee Medical Center, Loveland, Colorado
  - IACT Health, Columbus, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Duke University Medical Center, Durham, North Carolina
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Gibbs Cancer Center & Research Institute, Spartanburg, South Carolina
  - Parkland Health and Hospital System, Dallas, Texas
  - The University of Texas Southwestern Medical Center, Dallas, Texas
  - Cancer Care Northwest, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Squillace S, Salvemini D. Nitroxidative stress in pain and opioid-induced adverse effects: therapeutic opportunities. Pain. 2022 Feb 1;163(2):205-213. doi: 10.1097/j.pain.0000000000002347. No abstract available. PMID 34145168

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1: Subjects in Phase 1 received 100mg of GC4711 by 15 min IV prior to each administration of SBRT. SBRT was administered as a dose of 10-12 Gy per fraction in a total of 5 fractions within 10 calendar days.
- Phase 2 Placebo +SBRT: Subjects in Phase 2 received Placebo by a 15 min IV prior to each administration of SBRT. SBRT was administered as a dose of 10-12 Gy per fraction in a total of 5 fractions within 10 calendar days.
- Phase 2 GC4711 +SBRT: Subjects in Phase 2 received 100mg of GC4711 by 15 min IV prior to each administration of SBRT. SBRT was administered as a dose of 10-12 Gy per fraction in a total of 5 fractions within 10 calendar days.
Period: Overall Study
Arm/Group | Phase 1 | Phase 2 Placebo +SBRT | Phase 2 GC4711 +SBRT
Started | 7 | 20 | 20
Completed | 6 | 1 | 1
Not Completed | 1 | 19 | 19
Not completed — Withdrawal by Subject | 1 | 0 | 0
Not completed — Death | 0 | 1 | 2
Not completed — Sponsor Terminated Study | 0 | 18 | 17

BASELINE CHARACTERISTICS:
Groups:
- Phase 2 Placebo +SBRT: Subjects in Phase 2 received 100mg of Placebo by 15 min IV prior to each administration of SBRT. SBRT was administered as a dose of 10-12 Gy per fraction in a total of 5 fractions within 10 calendar days.
- Total: Total of all reporting groups
Arm/Group | Phase 1 | Phase 2 Placebo +SBRT | Phase 2 GC4711 +SBRT | Total
Number analyzed (Participants) | 7 | 20 | 20 | 47
Age, Customized [Count of Participants; unit: Participants]
  < 65 | 3 | 7 | 3 | 13
  >/= 65 | 4 | 13 | 17 | 34
  65-74 | 2 | 7 | 9 | 18
  >/=75 | 2 | 6 | 8 | 16
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 7 | 19
  Male | 5 | 10 | 13 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 5 | 8
  White | 7 | 16 | 15 | 38
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients With a Complete Response or Partial In-field Tumor Response Based on the RECIST 1.1 Criteria Through 6 Months Following SBRT.
Description: Subjects were required to have a baseline CT (chest, abdomen, and pelvis) and then were re-assessed by the same imaging modality at 6 months, 12 months, 18 months, and 24 months following the administration of GC4711/Placebo +SBRT and compared to the previous best response using RECIST 1.1 criteria.
Time Frame: 6 months, 12 months, 18 months and 24 months post SBRT and GC4711+Placebo
Population: Intent to Treat population includes all subjects enrolled/randomized to the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1 | Phase 2 Placebo +SBRT | Phase 2 GC4711 +SBRT
Number analyzed (Participants) | 7 | 20 | 20
Participants
  CR-Complete Response | 0 | 0 | 1
  PR-Partial Response | 2 | 6 | 6
  SD-Stable Disease | 5 | 4 | 6
  PD-Progressive Disease | 0 | 0 | 0
  NE-Not Evaluable | 0 | 10 | 7

ADVERSE EVENTS:
Time Frame: All adverse events were collected from Day 1 of dosing with GC4711/Placebo +SBRT through 90 days post SBRT (Total of 3.5 months)
Arm/Group | Phase 1 | Phase 2 Placebo +SBRT | Phase 2 GC4711 +SBRT
All-Cause Mortality (participants affected / at risk) | 0/7 | 1/20 | 2/20
Serious Adverse Events (participants affected / at risk) | 1/7 | 1/20 | 1/20
Other Adverse Events (participants affected / at risk) | 7/7 | 20/20 | 19/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=7) | Phase 2 Placebo +SBRT (N=20) | Phase 2 GC4711 +SBRT (N=20)
Cardiac Arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Pericardial Effusion (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1 (N=7) | Phase 2 Placebo +SBRT (N=20) | Phase 2 GC4711 +SBRT (N=20)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Leuckocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Photopsia (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Retinal Vascular Disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 1 (1) | 2 (2)
Vision Impairment (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Vitreous floaters (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal Pain Lower (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 3 (3) | 3 (3) | 2 (2)
Dry Mouth (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 3 (3) | 1 (1)
Eructation (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Hypoaesthesia oral (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 5 (5) | 5 (5) | 9 (9)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Oesophageal disorder (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oral dysaesthesia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 3 (3) | 0 (0)
Axillary Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 0 (0) | 0 (0) | 1 (1)
Chills (General disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 6 (6) | 10 (10) | 11 (11)
Feeling Hot (General disorders) | 0 (0) | 0 (0) | 1 (1)
Gait Disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Discomfort (General disorders) | 0 (0) | 1 (1) | 1 (1)
Infusion Site Erythema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Infusion Site Pain (General disorders) | 1 (1) | 1 (1) | 1 (1)
Infusion Site Swelling (General disorders) | 1 (1) | 0 (0) | 0 (0)
Injection Site Pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Injection site reaction (General disorders) | 1 (1) | 0 (0) | 1 (1)
Localised Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0)
Non Cardiac Chest Pain (General disorders) | 2 (2) | 2 (2) | 2 (2)
Oedema Peripheral (General disorders) | 1 (1) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 2 (2) | 1 (1)
COVID 19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 3 (3)
Radiation Associated Pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation Skin Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Rib Fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Skin Laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Vaccination complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood Chloride decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Blood Chloride decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Blood Creatinine increased (Investigations) | 1 (1) | 1 (1) | 0 (0)
Glomerular filtration rate decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Heart Rate Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
High Density Lipoprotein decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
International Normalised ratio Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 1 (1) | 5 (5) | 1 (1)
Monocyte count Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count increased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Platelet Count Decreased (Investigations) | 0 (0) | 2 (2) | 0 (0)
Red Blood Cell Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Serum Ferritin Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Weight Decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
White Blood Cell Count Decreased (Investigations) | 0 (0) | 1 (1) | 1 (1)
White Blood Cell Increased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased Appetite (Metabolism and nutrition disorders) | 0 (0) | 3 (3) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Back Pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 2 (2) | 0 (0)
Flank Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Joint Stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Metatarsalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 0 (0)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 0 (0)
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 1 (1)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 1 (1)
Plantar Fasciitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (2) | 2 (2) | 8 (8)
Essential tremor (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 3 (3) | 4 (4)
Hypersomnia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Paraesthesia (Nervous system disorders) | 3 (3) | 0 (0) | 5 (5)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Sedation (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Taste Disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional State (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Glycosuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Proteinuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary Tract Obstruction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nipple Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 9 (9) | 5 (5)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 6 (6) | 1 (1)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 1 (1)
Pulmonary Fibrosis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 4 (4) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Night Sweats (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin Tightness (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Flushing (Vascular disorders) | 1 (1) | 0 (0) | 1 (1)
Hot Flash (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
Hypotension (Vascular disorders) | 3 (3) | 4 (4) | 4 (4)

LIMITATIONS AND CAVEATS:
Study was terminated early by the Sponsor based on a the results of a futility analysis that was conducted on another program and the Sponsor decided to terminate the develop of GC4711. The last randomized subject did not complete protocol therapy but was followed for safety for a period of 30 days post the last administration of GC4711/Placebo +SBRT.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-04-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT04476797/Prot_SAP_000.pdf